CLINICAL TRIAL: NCT04773548
Title: Feasibility and Safety of a Virtual-Reality Based Job Interview Training Tool in Teenagers With High-Functioning Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-1036-18
Record Dates: First submitted 2021-02-25; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR-JIT (Experimental)
  Interventions: Other: VR-JIT

INTERVENTIONS:
Other: VR-JIT — Job interview with virtual interviewer

SUMMARY:
The current project involves the application of a VR job training software. We propose to use an interactive VR job interview practice system, Virtual Reality Job Interview Training (VR-JIT), in youths with ASD at the highschool level. This system was developed to bolster job interview practice skills and to help reduce anxiety in adults with ASD. However, it has never before been used in individuals under the age of 18. Our hope is that if this program is utilized in individuals while they are still in highschool, we can target those persons before the window for which risk of unemployment appears to be highest for ASD youths, immediately after high school graduation.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 13 and 18
* Have a diagnosis of ASD or a typically developing child
* Be able to speak and read English fluently

Exclusion Criteria:

* I had a stroke, TBI, or neurologic injury or disease in the past
* I have a history of significant psychiatric illness (like bipolar, schizophrenia, or psychosis)
* I have uncontrolled seizures or other unstable medical complications

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2020-10-24 (Actual); Study Completion 2020-10-24 (Actual)

PRIMARY OUTCOMES:
Change in mock job interview | 7 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided